CLINICAL TRIAL: NCT06537505
Title: An Exploratory Clinical Study of Microwave Ablation Combined With Immunotherapy ± Anti-angiogenic Drugs in the Treatment of Advanced Second-line and Above Solid Tumors
Brief Title: A Study of Microwave Ablation Combined With Immunotherapy ± Anti-angiogenic Drugs in the Treatment of Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beidahuang Industry Group General Hospital (Other)
Responsible Party: Principal Investigator, LiuMingyang, Associate Chief Physician, Beidahuang Industry Group General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-HLJ-010
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microwave ablation combined with immunotherapy and anti-angiogenic drugs (Experimental): microwave ablation combined with adebrelimab and apatinib
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Procedure: microwave ablation
- microwave ablation combined with immunotherapy (Experimental): microwave ablation combined with adebrelimab
  Interventions: Drug: Adebrelimab; Procedure: microwave ablation

INTERVENTIONS:
Drug: Adebrelimab — Q3W,IV
  Other Names: SHR-1316
Drug: Apatinib — QoD
  Arms: microwave ablation combined with immunotherapy and anti-angiogenic drugs
Procedure: microwave ablation — microwave ablation

SUMMARY:
This is a multi-center, phase Il trial to evaluate the efficacy and safety of microwave ablation combined with immunotherapy ± anti-angiogenic drugs in the treatment of advanced second-line and above solid tumors.

DETAILED DESCRIPTION:
This study plans to recruit 60 patients witha dvanced second-line and above solid tumors observe and evaluate the effectiveness and safety of microwave ablation combined with immunotherapy ± anti-angiogenic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically confirmed advanced non-small cell lung cancer or hepatocellular carcinoma;
2. Previously received systemic treatment;
3. Expected survival period > 3 months;
4. Age: 18-75 years old, male or female;
5. ECOG PS: 0-2 points;
6. The function of important organs meets the following requirements: a) Absolute neutrophil count ≥1.5×109/L, platelet ≥90×109/L, hemoglobin ≥90g/dL; b) Bilirubin ≤3 times ULN (patients drained by retrograde technique can be included); ALT and AST ≤5 times ULN, albumin>35g/ml, prothrombin time prolonged <6 seconds; c) Creatinine <120 μmol/L, or MDRD creatinine clearance >60 mL/min;
7. Women of childbearing age must have a negative pregnancy test (βHCG) before starting treatment, and women of childbearing age and men (having sexual relations with women of childbearing age) must agree to use effective contraceptive measures uninterruptedly during treatment and for 6 months after the last treatment dose;
8. The patient voluntarily joined this study and signed the informed consent form.

Exclusion Criteria:

1. Patients who have had other malignant tumors in the past or at the same time within 5 years, but excluding cured basal cell carcinoma of the skin, cervical carcinoma in situ, superficial or non-invasive bladder cancer, etc.
2. Patients with severe bleeding tendency and coagulation dysfunction that cannot be corrected in the short term;
3. Patients with severe pulmonary fibrosis and pulmonary hypertension;
4. Patients with infectious and radioactive inflammation around the lesion and skin infection at the puncture site that is not well controlled;
5. Systemic infection, high fever >38.5 ℃;
6. Severe anemia, dehydration and severe nutritional metabolism disorder that cannot be corrected or improved in a short period of time;
7. Poorly controlled malignant pleural effusion;
8. Uncontrolled, symptomatic brain metastasis or a history of difficult-to-control mental illness or severe intellectual or cognitive impairment;
9. Subjects with active, known or suspected autoimmune diseases, hypothyroidism that only requires hormone replacement therapy, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or alopecia) can be selected;
10. Congestive heart failure, uncontrollable arrhythmias, myocardial infarction within 6 months, unstable angina, stroke or transient ischemic attack;
11. Patients who cannot comply with the trial protocol or cannot cooperate with follow-up;
12. History of psychotropic drug abuse, alcoholism or drug abuse;
13. Human immunodeficiency virus (HIV, HIV 1/2 antibody) positive;
14. Those who are considered by the researchers to be unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 24 months
  Determined using RECIST V1.1 criteria, defined as best overall response (CR or PR)

SECONDARY OUTCOMES:
Disease control rate | up to 24 months
  Disease Control Rate determined usina RECIST V1.1 criteria.
Progression-free Survival | up to 36 months
  Defined as the time from randomization to the first occurrence of disease progression
Overall Survival | up to 36 months
  Defined as the time from randomization to death from any cause.
incidence rate of AE | up to 36 months
  Incidence, nature, and severity of adverse events graded according to the NCI CCAE

OTHER OUTCOMES:
explore immune resistance mechanisms | up to 36 months
  to explore immune resistance mechanisms

IPD SHARING:
Plan to Share IPD: No